CLINICAL TRIAL: NCT05712564
Title: Observational Survey on Fatigue Levels in Relation to Depressive Disorders and Insomnia in Adult Patients with Marfan Syndrome and Hypermobile Ehlers-Danlos Syndrome
Brief Title: Fatigue, Depressive Disorders and Insomnia in Adult Patients with Marfan Syndrome and Ehlers-Danlos Syndrome: Survey
Acronym: FAMED
Status: Completed | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Alessandro Pini, Principal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: FAMED
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Rare Diseases; Fatigue; Insomnia; Depression
Keywords: Marfan syndrome; Ehlers-Danlos syndrome; Fatigue; Survey
MeSH Terms: conditions — Rare Diseases; Fatigue; Sleep Initiation and Maintenance Disorders; Depression; Marfan Syndrome; Ehlers-Danlos Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MFS_cohort: Adult patients with Marfan syndrome
  Interventions: Other: Questionnaire
- hEDS_cohort: Adult patients with hypermobile Ehlers-Danlos syndrome
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire for fatigue assessment

SUMMARY:
The goal of this observational study is to describe and assess the presence of perceived fatigue in subjects with MFS and EDS. the main question it aims to answer through the FSS instrument is:

* The relationship of fatigue with physical and psychological characteristics, the presence of depressive disorders and insomnia.

DETAILED DESCRIPTION:
Marfan syndrome (MFS) and hypermobile Ehlers-Danlos Syndrome (hEDS) are rare diseases of the connective tissue presenting peculiar symptoms as well as high mortality due to complications related to dilatation and dissection of the ascending aorta and great arteries. Life expectancy of patients with MFS and hEDS has improved markedly in the last decades, but still remains lower than that of the general population. Fatigue represent one of the main causes that limit the quality of life in these populations. The Fatigue Severity Scale (FSS) is a questionnaire widely used in populations with chronic diseases and has been previously applied in MFS and hEDS population: indeed, fatigue interferes with activities of daily living and the presence of chronic pain. However, the potential correlations that fatigue may have with different aspects of psychological well-being (i.e. insomnia and depression) were not investigated in MFS and hEDS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 or greater with clinical and/or genetic diagnosis of Marfan syndrome;
* Subjects aged 18 or greater with clinical and/or genetic diagnosis of hypermobile Ehlers-Danlos syndrome;
* Signed informed consent;
* Ability to speak, read and write in Italian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollment of 200 subjects with MFS and hEDS currently in follow-up at the Cardiovascular Genetic Centre, IRCCS Policlinico San Donato. The study includes the involvement of subjects with hEDS currently in follow-up at Fondazione Ca' Granda IRCCS Policliclinico.
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Physical and psychological features | 10 months
  The mean, median, standard deviation and interquartile range will be used for continuous variables, whereas frequency and percentage will be applied for nominal and categorical variables. The Shapiro-Wilks test will be used to assess the Gaussian distributions.

SECONDARY OUTCOMES:
Psychosocial variables | 10 months
  The bivariate correlation analysis will be performed by calculating the Pearson or Spearman correlation coefficient

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Lombardy, Italy

REFERENCES:
- [Derived] Udugampolage N, Taurino J, Bassotti A, Pini A, Caruso R, Callus E, Magon A, Conte G, De Angeli G, Paglione G, Baroni I, Trifiro G. Exploring fatigue in Marfan and hypermobile Ehlers-Danlos syndromes: an analytical cross-sectional study in two Italian healthcare centres. BMJ Open. 2025 Jan 6;15(1):e087298. doi: 10.1136/bmjopen-2024-087298. PMID 39762099